CLINICAL TRIAL: NCT06611852
Title: Efficacy of Combined Interferential Therapy and Electronic Cupping Therapy for Chronic Constipation Management
Acronym: Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Middle East University (Other)
Responsible Party: Principal Investigator, Emad Eldin Mohamed, assistant professor, Middle East University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2513; middle east university (Other: middle east university)
Record Dates: First submitted 2024-09-18; First posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Constipation
Keywords: Chronic Constipation; Interferential Therapy; Electronic Cupping Therapy
MeSH Terms: conditions — Constipation | interventions — Exercise; Population Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Group (A) (Experimental): received aerobic exercises
  Interventions: Other: Aerobic exercise
- Group (B) (Experimental): received electronic cupping therapy
  Interventions: Other: electronic cupping therapy in addition to aerobic exercise
- Group (C) (Experimental): received interferential therapy
  Interventions: Other: interferential therapy in addition to aerobic exercise
- Group (D) (Experimental)
  Interventions: Other: interferential therapy, electronic cupping therapy in addition to aerobic exercises

INTERVENTIONS:
Other: Aerobic exercise — Warm-up (5 minutes): Started with a 5-minute warm-up on the stationary bike at a low intensity to prepare the muscles for the workout.
  Interval Training (15 minutes): Alternated between 1 minute of high-intensity cycling (pedaling at a faster pace with higher resistance) and 2 minutes of moderate-intensity cycling (steady pace with moderate resistance). This interval was repeated for a total of 15 minutes.
  Hill Climbing (10 minutes): The resistance was increased on the stationary bike to simulate climbing a hill. Pedal at a slower pace but with higher resistance for 10 minutes to engage the muscles of legs and core.
  Cool Down (5 minutes): The stationary cycling session was finished with a 5-minute cool down at a low intensity to gradually lower the heart rate and avoid fatigue.
  Other Names: Group (A)
  Arms: Group (A)
Other: electronic cupping therapy in addition to aerobic exercise — Four devices of electronic cupping therapy were equipped with 3.5-inch diameter cups (Becommend, model number: BE007, ASIN: B09PVF72RJ, China).
  Arms: Group (B)
Other: interferential therapy in addition to aerobic exercise — interferential current (Endomed 482, SN/29.382, Netherlands) was delivered by the following parameters: a carrier frequency of 5-kHz, a beat frequency of 80-160 Hz, and an intensity level below 33 mA. Four carbon rubber electrodes (8x12 cm) were used and fixed by a large abdominal strap with a wet spongy
  Arms: Group (C)
Other: interferential therapy, electronic cupping therapy in addition to aerobic exercises — interferential therapy, electronic cupping therapy in addition to aerobic exercises
  Arms: Group (D)

SUMMARY:
Constipation is a common gastrointestinal issue affecting individuals worldwide. Interferential therapy, a form of electrotherapy, has been suggested to have potential benefits in improving gastrointestinal motility and relieving constipation symptoms. Introducing of a new method like electronic cupping therapy with interferential therapy may optimize the therapeutic outcomes by potentially increasing bowel movements and improving overall gastrointestinal function.

DETAILED DESCRIPTION:
Objective: The purpose of this study was to assess the effectiveness of a combined treatment regimen that includes interferential therapy and electronic cupping therapy on the symptoms of chronic constipation, as well as gastrointestinal health outcomes.

Methods: This study involved 110 patients with chronic constipation, consisting of 60 females and 50 males, ranging in age from 20 to 40 years. Each participant underwent evaluations using Abdominal Ultrasonography and a standardized constipation scoring system. All participants were allocated into three groups; Group (A) received interferential therapy with aerobic exercises, Group (B) received electronic cupping therapy and aerobic exercise in the form of treadmill exercise and stationary bicycle 3 sessions/week for four weeks, and Group (c) received interferential therapy, electronic cupping therapy in addition to aerobic exercises.

ELIGIBILITY:
Inclusion Criteria:

* history of Chronic Constipation (CC), as defined by either experiencing two or fewer Complete Spontaneous Bowel Movements (CSBMs) per week for a minimum of 6 consecutive months before the screening visit
* Reporting a sensation of incomplete evacuation or straining during at least a quarter of their bowel movements (according to the generally accepted definition of constipation).
* Patients must have had CC persisting for more than 6 months, failed to respond to or be intolerant of medical treatment for at least 3 months

Exclusion Criteria:

* pregnant or lactating women
* Chronic Constipation (CC) resulting from anorectal malformations such as colorectal or anal organic lesions, pelvic floor disorders requiring surgical intervention as determined by the investigator (such as rectal prolapse, rectocele, or enterocele)
* presence of implanted electronic devices like cardiac pacemakers, defibrillators, cardiac pumps, or spinal stimulators
* CC attributable to medications or neurologic, endocrine, or metabolic conditions
* prior history of partial colectomy; conditions like megacolon, megarectum, or colonic inertia
* skin abnormalities that hinder the placement of electrodes
* women lacking adequate contraception (hormonal or intrauterine device).

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-10-20 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Ultrasonography | 6 weeks
  Ultrasonography (M-Turbo, Sonosite, Bothell, WA, USA) was used to assess the large intestine during CC by using imaging technology that gave the healthcare professionals the ability to visualize the structure and function of the patients' bowel with a curved-array (2-5 MHz) probe.
Constipation scoring system. | 6 weeks
  A constipation scoring system was used to evaluate the severity of CC. It measures the frequency of the bowel movements, stool consistency, straining during defecation, and sensation of incomplete evacuation. It produces a numerical score ranging from 0 to 30, with 0 indicating no constipation and 30 indicating severe constipation

CONTACTS AND LOCATIONS:
Locations (1):
- October 6 university, October City, Giza Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No